CLINICAL TRIAL: NCT01516190
Title: The Preoperative Health & Body Study
Acronym: PreHab
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Yale University (Other); Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-182
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: stage I-III breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Group (Active Comparator): Supervised exercise sessions and independent exercise
  Interventions: Behavioral: Exercise
- Mind-Body Group (Active Comparator): Surgical preparation program
  Interventions: Behavioral: Surgical preparation program

INTERVENTIONS:
Behavioral: Exercise — Supervised exercise sessions and independent exercise
  Arms: Exercise Group
Behavioral: Surgical preparation program — Book, tapes, CD
  Arms: Mind-Body Group

SUMMARY:
This study is designed to look at the changes that occur in women who take part in exercise and Mind-Body programs between breast cancer diagnosis and breast surgery. The investigators will look at changes in stress, anxiety, mood and quality of life, to see if these types of short programs can make women feel better during this time. The investigators are also interested in looking at whether a short exercise or Mind-Body program leads to any changes in markers in breast cancer cells, such as their growth and death rates, or in blood hormones such as insulin, which have been linked to breast cancer development.

Since the investigators do not know if these blood or tumor tests have any relationship to cancer recurrence, the investigators do not plan to share the results of these tests with you or your physician.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically confirmed stage I-III breast cancer
* Planning to undergo definitive surgical management with lumpectomy or mastectomy with in the next 8 weeks.
* Willing and able to participate in the intervention for at least 3 weeks prior to surgery.
* ECOG performance status of 0 or 1
* Approval by oncologist or surgeon
* Willingness to be randomized.
* English speaking and able to read English

Exclusion Criteria:

* Concurrent other malignancy or history of other malignancy treated within the past 3 years (other than non-melanoma skin cancer or in situ cervical cancer)
* Presence of metastatic disease
* Scheduled to receive any form of neoadjuvant cancer therapy
* Locally advanced breast cancer not amenable to primary surgery
* History of prior ipsilateral breast cancer
* Taking tamoxifen, raloxifene or an aromatase inhibitor at the time of breast cancer diagnosis
* Absolute contraindications to maximal exercise testing as recommended by the American Thoracic Society
* Any condition which in the investigator's opinion makes the subject unsuitable for study participation
* Participating in another clinical study with competing study outcomes
* Pregnant (i.e., positive beta-HCG) or breast feeding
* Unable to comply with protocol and/or not available for follow-up assessments
* Participation in more than 90 minutes a week of moderate-intensity recreational activity (not including activities such as gardening, bowling, golfing with a cart) as assessed by the Leisure Score Index of Godin Leisure- Time Exercise Questionnaire (LSI) (Appendix I) or recent participation (past 6 months) in two or more strength training sessions per week.
* Diabetes mellitus requiring insulin or oral agents; patients with diet-controlled diabetes will be allowed to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Impact of Exercise on Ki-67 | 3 years
  To explore the impact of exercise upon Ki-67, a tissue-based biomarker associated with breast cancer risk and progression.
Feasibility of intervention in women with newly diagnosed breast cancer | 3 years
  To evaluate the feasibility of conducting a window of opportunity study utilizing exercise and mind-body intervention in women with newly diagnosed breast cancer

SECONDARY OUTCOMES:
Impact of exercise on biomarkers | 3 years
  To evaluate the impact of a 3-6 week intensive exercise intervention upon concentrations of serum matabolic and inflammatory biomarkers (insulin, glucose, IGF-1, IGFBP's, IL-2, IL-6, CRP, TNFa)
Impact of exercise on receptors | 3 years
  To explore the impact of a 3-6 week exercise intervention upon expression of metabolic, sex steroid and related receptors in malignant breast tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Knoerl R, Giobbie-Hurder A, Sannes TS, Chagpar AB, Dillon D, Dominici LS, Frank ES, Golshan M, McTiernan A, Rhei E, Tolaney SM, Winer EP, Yung RL, Irwin ML, Ligibel JA. Exploring the impact of exercise and mind-body prehabilitation interventions on physical and psychological outcomes in women undergoing breast cancer surgery. Support Care Cancer. 2022 Mar;30(3):2027-2036. doi: 10.1007/s00520-021-06617-8. Epub 2021 Oct 14. PMID 34648061